CLINICAL TRIAL: NCT03044496
Title: Near-infrared Spectroscopy to Assess Changes in Tissue Oxygenation Following Supraclavicular Plexus Block in Patients Undergoing Vascular Surgery
Brief Title: NIRS Measurement After SCP Block
Status: Completed | Type: Observational
Sponsor: Marienhospital Stuttgart (Other)
Responsible Party: Principal Investigator, Dr. Christoph Ilies, Principal Investigator, Assistant Medical Director Dpt. for Anaesthesiology, Marienhospital Stuttgart
Other Study IDs: NIRS after SCP block
Record Dates: First submitted 2017-01-31; First posted 2017-02-07 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Arterio-venous Fistula
Keywords: NIR Spectroscopy; Nerve Blockade; Surgical Arteriovenous Shunt
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Supraclavicular Nerve Block: Patients undergoing vascular surgery for creation or revision of an arterio-venous fistula. Intervention: supraclavicular plexus block for anaesthesia. NIRS measurement before and after brachial plexus block.
  Interventions: Drug: Supraclavicular nerve block

INTERVENTIONS:
Drug: Supraclavicular nerve block — Supraclavicular nerve block using ultrasound and 10ml ropivacaine 0.5% with 20ml mepivacaine 1%

SUMMARY:
Peripheral regional anesthesia induces a sympathectomy-like effect with neurovascular changes causing increased arterial blood flow and venodilatation .

Near-infrared spectroscopy (NIRS) can be applied to different kinds of tissue providing oxygen saturation by detecting the absorption and reflection of near-infrared light .

The effect on peripheral tissue oxygenation in patients undergoing arteriovenous fistula revision has not yet been examined. We postulate an increase in tissue oxygenation by sympathicolysis caused by peripheral regional anesthesia that might be the reason for beneficial outcome. The aim of our study was to demonstrate the effect of a supraclavicular plexus block in this group of patients.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing surgery under regional anaesthesia

Exclusion Criteria:

* patients refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing shunt surgery under supraclavicular plexus block
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
NIRS after block | 5 minutes before block until 30 minutes after block
  Absolute change from baseline value in tissue oxygenation

SECONDARY OUTCOMES:
Difference between both arms | 5 minutes before block until 30 minutes after block
  Absolute difference in tissue oxygenation between blocked arm and contralateral arm

CONTACTS AND LOCATIONS:
Locations (1):
- Marienhospital Stuttgart, Dpt. of Anaesthesiology, Stuttgart, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Keuler J, Weiss C, Klemm K, Pochhammer J, Schmidt R, Ilies C. Assessing changes in tissue oxygenation by near-infrared spectroscopy following brachial plexus block for arteriovenous fistula surgery: A prospective observational pilot study. Eur J Anaesthesiol. 2018 Oct;35(10):759-765. doi: 10.1097/EJA.0000000000000871. PMID 30124502